CLINICAL TRIAL: NCT00192348
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety and Tolerability of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold Adapted (CAIV-T) in Healthy Infants
Brief Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety and Tolerability of Influenza Virus Vaccine,(CAIV-T) in Healthy Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D153-P518
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2006-10

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
Trial to compare the safety and tolerability of one and two doses of influenza virus vaccine.

DETAILED DESCRIPTION:
The objective of this study was to compare the safety and tolerability of one and two doses of influenza virus vaccine, trivalent, types A and B, live cold-adapted liquid (CAIV-T) with placebo when administered intranasally to healthy infants aged 6 < 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* children at least 6 weeks of age and less than 24 weeks of age at the time of enrollment, of >37 weeks gestational age and with a birth weight of >2500 g, and in good health as determined by medical history, physical examination and clinical judgment;
* whose parent/legal guardian provided written informed consent after the nature of the study was explained;
* who, along with their parent or legal guardian, were available for the three month duration of the trial (from enrollment to study completion);
* whose parent(s)/legal guardian(s), could be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria:

* whose parents or legal guardians were perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents;
* who received any blood products, including immunoglobulin, in the period from birth through to the conclusion of the study;
* had an immunosuppressed or an immunocompromised individual living in the same household;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccines or placebo;
* who were administered any live virus vaccine within one month prior to enrollment; or expected to receive another live vaccine within 1 month of vaccination in the study.
* for whom there was intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* who received a dose of influenza treatment (commercial or investigational) two weeks prior to enrollment. The prophylactic use of influenza antivirals was not permitted;
* who, at anytime prior to study enrollment, received any influenza vaccine (commercial or investigational);
* with a respiratory illness with wheezing within two weeks prior to each dose of study vaccine;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use was anticipated during the study;
* with any medical conditions that in the opinion of the investigator might have interfered with interpretation of the study results.

Note: Pregnancy in any person who had regular contact with the subjects was not considered a contraindication to enrollment.

Ages: 6 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2002-05; Study Completion 2002-12

PRIMARY OUTCOMES:
- To compare the safety and tolerability of one and two doses of influenza virus vaccine, trivalent,(CAIV-T) with placebo when administered intranasally

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- University of Tampere, Tampere, Finland

REFERENCES:
- [Derived] Vesikari T, Karvonen A, Smith HM, Dunning A, Razmpour A, Saville MK, Gruber WC, Forrest BD. Safety and tolerability of cold-adapted influenza vaccine, trivalent, in infants younger than 6 months of age. Pediatrics. 2008 Mar;121(3):e568-73. doi: 10.1542/peds.2007-1405. Epub 2008 Feb 25. PMID 18299305